CLINICAL TRIAL: NCT03754842
Title: Effect of Nicotinamide Riboside and Pterostilbene Supplementation on Muscle Regeneration in Elderly Humans - A Randomized, Placebo-controlled, Clinical Trial
Brief Title: Effect of Nicotinamide Riboside and Pterostilbene Supplementation on Muscle Regeneration in Elderly Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AU2018-11-19
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-03

CONDITIONS: Muscle Injury
MeSH Terms: interventions — nicotinamide-beta-riboside; Pterocarpus marsupium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo (twice daily)
- Nicotinamide Riboside + Pterostilbene (Experimental)
  Interventions: Other: Nicotinamide Riboside/Pterostilbene (500 mg/100 mg twice daily)

INTERVENTIONS:
Other: Placebo (twice daily) — Matching placebo
  Arms: Placebo
Other: Nicotinamide Riboside/Pterostilbene (500 mg/100 mg twice daily) — Elysium Basis TM, Elysium Health, Inc., NY, USA
  Arms: Nicotinamide Riboside + Pterostilbene

SUMMARY:
Successful skeletal muscle regeneration depends on a functional pool of muscle stem cells, termed satellite cells (SC). SC are in a quiescent state throughout adulthood, but undergo multiple cycles of proliferation and self-renewal in response to muscle damage. During aging, there is a loss of SC quiescence, and SC more readily enter an ageing-state impairing their function.

Animal studies have revealed a common denominator for increasing SC function and activity, namely Sirtuin activation. Natural stimulators of Sirtuins includes Nicotinamide Riboside (NR) (a Nicotinamide adenine dinucleotide (NAD+) precursor) and the polyphenol Pterostilbene (PT). In this study, we aim to investigate if NR+PT supplementation will promote skeletal muscle regeneration after muscle damage in elderly humans by enhanced recruitment of SC.

DETAILED DESCRIPTION:
14 days after start of placebo or NR/PT (500/100 mg twice daily) supplementation a muscle damage will induced in the m. vastus lat. by electric stimulation combined with eccentric work in a dynamometer. Muscle biopsies will be collected at 2 hours, 2, 8 and 30 days post damage and placebo or NR/PT supplementation will continue for the whole study period (45 days).

ELIGIBILITY:
Inclusion Criteria:

* Written signed consent
* Age: 55-80
* BMI: 20-28 (kg/(m2))
* Non-smoker

Exclusion Criteria:

* Endocrine disease, neurological or muscle disease
* Other severe disease
* High daily activity level (>30 min / day)

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Presence of Satellite Cells | Change from baseline up to 45 days
  quantified by immunohistochemistry in muscle biopsies

SECONDARY OUTCOMES:
Activation of Satellite cells | Change from baseline up to 45 days
  determined by immunohistochemistry and FACS
Presence of macrophages | Change from baseline up to 45 days
  determined by immunohistochemistry and FACS
Presence of Fibro/Adipogenic Progenitors | Change from baseline up to 45 days
  quantified by FACS
Presence of damaged muscle fibers | Change from baseline up to 45 days
  determined by immunohistochemistry
Presence of muscle regenerative fibers | Change from baseline up to 45 days
  determined by immunohistochemistry
Presence of autophagy in relation to muscle damage | Change from baseline up to 45 days
  determined by Western blot and PCR
Lipid accumulation in skeletal muscle tissue and liver | Change from baseline to 8 days
  determined by magnetic resonance spectroscopy
Blood glucose response in relation to muscle damage | Change from baseline to 8 days
  determined by Continuous glucose monitoring
Body composition (lean body mass and fat body mass) | Change from baseline to 45 days
  measured by Dual energy X-ray absorptiometry
Muscle strength | Change from baseline up to 45 days
  determined from maximal voluntary contraction of the m. quadriceps femoris

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jensen JB, Dollerup OL, Moller AB, Billeskov TB, Dalbram E, Chubanava S, Damgaard MV, Dellinger RW, Trost K, Moritz T, Ringgaard S, Moller N, Treebak JT, Farup J, Jessen N. A randomized placebo-controlled trial of nicotinamide riboside and pterostilbene supplementation in experimental muscle injury in elderly individuals. JCI Insight. 2022 Oct 10;7(19):e158314. doi: 10.1172/jci.insight.158314. PMID 35998039